CLINICAL TRIAL: NCT00876109
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating Two Dosing Schedules of PI3-Kinase Inhibitor (GDC-0941) in Patients With Locally Advanced or Metastatic Solid Tumors for Which Standard Therapy Either Does Not Exist or Has Proven Ineffective or Intolerable
Brief Title: A Study of GDC-0941 in Participants With Locally Advanced or Metastatic Solid Tumors for Which Standard Therapy Either Does Not Exist or Has Proven Ineffective or Intolerable
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GDC4255g; GO01300 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-03-13; First posted 2009-04-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
Keywords: Metastatic Solid Tumors; PI3K; PI3K Inhibitors
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

ARMS (3):
- Group A: GDC-0941 QD Dose Escalation (Experimental): Participants will receive GDC-0941 for up to 1 year, administered orally QD at a starting dose of 15 milligrams (mg).
  Interventions: Drug: GDC-0941
- Group B: GDC-0941 BID Dose Escalation (Experimental): Participants will receive GDC-0941 for up to 1 year, administered orally BID at a starting dose determined from Group A assessments.
  Interventions: Drug: GDC-0941
- Group C: GDC-0941 QD or BID Expansion (Experimental): Participants will receive GDC-0941 for up to 1 year, administered orally QD or BID. The dose/regimen will be determined on the basis of data from Groups A and B.
  Interventions: Drug: GDC-0941

INTERVENTIONS:
Drug: GDC-0941 — GDC-0941 will be administered in escalating oral doses QD or BID in Groups A and B, respectively. In Group C, the dose/regimen will be determined on the basis of data from Groups A and B. The overall starting dose will be 15 mg administered in the first cohort enrolled in Group A.
  Other Names: PI3-Kinase Inhibitor

SUMMARY:
This is an open-label, multicenter, Phase I, dose-escalation study to assess the safety, tolerability, and pharmacokinetics of orally administered GDC-0941 administered once daily (QD) and twice daily (BID) in the treatment of advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically documented, incurable, locally advanced or metastatic solid malignancy that has progressed or failed to respond to at least one prior regimen, and who are not candidates for regimens known to provide clinical benefit
* Evaluable or measurable disease per RECIST
* Life expectancy of greater than or equal to (>/=) 12 weeks
* Documented willingness to use an effective means of contraception (for both men and women) while participating in the study

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current malignancy
* History of Type 1 or 2 diabetes mellitus requiring regular medication
* Any condition requiring anticoagulants, such as warfarin, heparin, or thrombolytics
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known untreated central nervous system (CNS) malignancies or treated brain metastases that are not radiographically stable for >/=3 months
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Uncontrolled ascites requiring weekly large-volume paracentesis for 3 consecutive weeks prior to enrollment
* Active infection requiring intravenous (IV) antibiotics
* Requirement for any daily supplemental oxygen
* Uncontrolled hypomagnesemia or hypokalemia, defined as values below the lower limit of normal (LLN), or hypercalcemia above the upper limit of normal (ULN) for the institution despite adequate electrolyte supplementation or management
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the participant at high risk from treatment complications
* Significant traumatic injury within 3 weeks before Day 1
* Major surgical procedure within 4 weeks prior to initiation of study treatment
* Treatment with chemotherapy, hormonal therapy (except gonadotropin releasing hormone [GnRH] agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, or radiation therapy (except palliative radiation to bony metastases) as cancer therapy within 4 weeks prior to initiation of study treatment
* Palliative radiation to bony metastases within 2 weeks prior to initiation of study treatment
* Need for chronic corticosteroid therapy for greater than (>) 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-10; Primary Completion 2012-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of GDC-0941 | Pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72 h) Day 1; pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24 h) Days 8 and 15; pre-dose (5 min) Days 22, 29, 36, and end of Cycles 1 to 12 (up to 1 year overall)
Terminal Elimination Half-Life (t1/2) of GDC-0941 | Pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72 h) Day 1; pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24 h) Days 8 and 15; pre-dose (5 min) Days 22, 29, 36, and end of Cycles 1 to 12 (up to 1 year overall)
Area Under the Concentration-Time Curve (AUC) of GDC-0941 | Pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72 h) Day 1; pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24 h) Days 8 and 15; pre-dose (5 min) Days 22, 29, 36, and end of Cycles 1 to 12 (up to 1 year overall)
Percentage of Participants with Adverse Events | Visits during treatment on Days 1, 2, 3, 4, 8, 15, 22, 29, 36; weekly during Cycle 2; every two weeks during Cycles 3 to 6; every month during Cycles 7 to 12; and up to 30 days after last dose (up to 1 year overall)
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Visits during treatment on Days 1, 2, 3, 4, 8, 15, 22, 29, 36
Percentage of Participants with Grade 3 or 4 Abnormalities in Safety-Related Laboratory Parameters | Visits at Baseline and during treatment on Days 1, 8, 15, 22, 29, 36; weekly during Cycle 2; every two weeks during Cycles 3 to 6; every month during Cycles 7 to 12; and up to 30 days after last dose (up to 1 year overall)
Time of Maximum Observed Concentration (Tmax) of GDC-0941 | Pre-dose (5 minutes [min]) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72 hours [h]) Day 1; pre-dose (5 min) and post-dose (0.5, 1, 2, 3, 4, 8, 12, 24 h) Days 8 and 15; pre-dose (5 min) Days 22, 29, 36, and end of Cycles 1 to 12 (up to 1 year overall)

SECONDARY OUTCOMES:
Duration of Objective Response According to RECIST | Tumor assessments as Baseline, Day 36, and every 8 weeks thereafter through Cycle 12 (up to 1 year overall)
Progression-Free Survival (PFS) According to RECIST | Tumor assessments as Baseline, Day 36, and every 8 weeks thereafter through Cycle 12 (up to 1 year overall)
Percentage of Participants by Best Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST) | Tumor assessments as Baseline, Day 36, and every 8 weeks thereafter through Cycle 12 (up to 1 year overall)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Hsu, M.D., Study Director — Genentech, Inc.
Locations (3):
- United States (3):
  - Scottsdale, Arizona
  - Boston, Massachusetts
  - Detroit, Michigan